CLINICAL TRIAL: NCT07268794
Title: A Multicenter, Prospective, Randomized Controlled Phase II Clinical Trial of Prostatectomy After Conversion Therapy With Second-generation Antiandrogen Agents Plus ADT in Patients With High-volume mHSPC(CONVERT-HB1)
Brief Title: CONVERT-HB1: Radical Prostatectomy After Systemic Therapy for High-volume Metastatic Hormone-sensitive Prostate Cancer
Acronym: CONVERT-HB1
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Ding-Wei Ye, Fudan University Shanghai Cancer Center (Fudan University Shanghai Cancer Hospital), Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MNWKQXJ20251102
Record Dates: First submitted 2025-11-16; First posted 2025-12-08 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-11

CONDITIONS: Metastatic Prostate Cancer; Prostate Cancer (Adenocarcinoma); Metastatic Hormone-Sensitive Prostate Cancer (mHSPC)
Keywords: High-volume mHSPC; Androgen deprivation therapy; Second-generation antiandrogens; Rezvilutamide; Radical prostatectomy; Radiotherapy; Conversion therapy
MeSH Terms: conditions — Prostatic Neoplasms; Adenocarcinoma | interventions — Androgen Antagonists; Docetaxel; Poly(ADP-ribose) Polymerase Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Systemic Therapy Alone (Active Comparator): Participants with high-volume metastatic hormone-sensitive prostate cancer (mHSPC) who achieve "conversion success" after induction systemic therapy will be randomized to this arm at either the 6-month or 12-month evaluation. Conversion success is defined based on PSMA PET/CT as all metastatic lesions showing no obvious uptake (SUVmax lower than liver SUVmean or blood pool SUVmean) and fulfilling all predefined clinical and radiological criteria for randomization.
  Patients randomized to Arm A will continue standard systemic therapy alone without local prostate surgery or radiotherapy. Systemic therapy consists of androgen deprivation therapy (ADT) using LHRH agonists or antagonists (e.g., goserelin, leuprolide, triptorelin, degarelix) combined with second-generation androgen receptor signaling inhibitors (such as rezvilutamide, enzalutamide, apalutamide, darolutamide, or abiraterone), with or without docetaxel and other systemic agents (e.g., PARP inhibitors such as olaparib), admini
  Interventions: Drug: Androgen Deprivation Therapy (ADT); Drug: Docetaxel; Drug: PARP Inhibitors and Other Systemic Agents
- Systemic Therapy Plus Local Prostate Treatment (Arm B) (Experimental): Participants with high-volume metastatic hormone-sensitive prostate cancer (mHSPC) who achieve "conversion success" after induction systemic therapy will be randomized to this arm at either the 6-month or 12-month evaluation. Conversion success is defined based on PSMA PET/CT as all metastatic lesions showing no obvious uptake (SUVmax lower than liver SUVmean or blood pool SUVmean) and fulfilling all predefined clinical and radiological criteria for randomization.
  Patients randomized to Arm B will receive local prostate treatment in addition to continued standard systemic therapy. Systemic therapy consists of ADT using LHRH agonists or antagonists (e.g., goserelin, leuprolide, triptorelin, degarelix) combined with second-generation androgen receptor signaling inhibitors (such as rezvilutamide, enzalutamide, apalutamide, darolutamide, or abiraterone), with or without docetaxel and other systemic agents (e.g., PARP inhibitors such as olaparib), administered according to approved labels
  Interventions: Drug: Androgen Deprivation Therapy (ADT); Drug: Docetaxel; Drug: PARP Inhibitors and Other Systemic Agents; Procedure: Radical Prostatectomy; Radiation: Prostate Radiotherapy

INTERVENTIONS:
Drug: Androgen Deprivation Therapy (ADT) — Androgen deprivation therapy using LHRH agonists or antagonists (e.g., goserelin, leuprolide, triptorelin, degarelix) according to local prescribing information and CSCO guideline recommendations. The specific drug, dose, and schedule are determined by the investigator and may be adjusted based on tolerability and adverse events.
Drug: Docetaxel — Intravenous docetaxel may be combined with ADT plus second-generation ARSis in selected patients according to contemporary guideline recommendations and investigator judgment. Dose and schedule follow approved labels and may be modified based on toxicity and tolerability.
Drug: PARP Inhibitors and Other Systemic Agents — Other systemic agents, including PARP inhibitors such as olaparib, may be used in combination with ADT and second-generation ARSis according to approved indications, molecular testing results, guideline recommendations, and investigator judgment.
Procedure: Radical Prostatectomy — Radical prostatectomy with bilateral seminal vesicle removal and, when appropriate, pelvic lymph node dissection, performed by experienced urologic surgeons via open, laparoscopic, or robot-assisted approach, in patients randomized to Arm B who have achieved conversion success on PSMA PET/CT
  Arms: Systemic Therapy Plus Local Prostate Treatment (Arm B)
Radiation: Prostate Radiotherapy — Definitive external-beam radiotherapy to the prostate delivered according to institutional standards and guideline recommendations, as an alternative local prostate treatment for patients randomized to Arm B who have achieved conversion success on PSMA PET/CT and are not undergoing radical prostatectomy
  Arms: Systemic Therapy Plus Local Prostate Treatment (Arm B)

SUMMARY:
This is a prospective, randomized, open-label, phase II multicenter clinical trial evaluating the efficacy and safety of radical prostatectomy in patients with high-volume metastatic hormone-sensitive prostate cancer (mHSPC) who achieve good response after systemic therapy with androgen deprivation therapy (ADT) plus second-generation antiandrogens such as rezvilutamide. All eligible patients will receive 6 months of induction systemic therapy (ADT plus second-generation androgen receptor signaling inhibitors, with or without docetaxel or other systemic agents). Patients who achieve PSMA PET/CT "conversion success" (no metabolically active lesions; all metastases with SUVmax below liver background or blood pool) will be randomized 1:1 to continue systemic therapy alone (control arm) or receive local prostate treatment (radical prostatectomy or radiotherapy) plus systemic therapy (experimental arm). The primary endpoint is radiographic progression-free survival (rPFS). Key secondary endpoints include overall survival (OS), biochemical progression-free survival (bPFS), PSA response rate, quality of life, conversion success rate, and safety.

ELIGIBILITY:
Inclusion Criteria:

1. Male patients aged >18 and ≤70 years, or with an estimated life expectancy >10 years.
2. Histologically or cytologically confirmed prostate adenocarcinoma with neuroendocrine differentiation ≤10%, and no small cell or signet-ring cell carcinoma component.
3. High-volume metastatic disease according to CHAARTED definition: presence of visceral metastasis and/or ≥4 bone lesions with at least one lesion outside the axial skeleton (vertebral bodies and pelvis).
4. Newly diagnosed metastatic hormone-sensitive prostate cancer (mHSPC) who started intensified endocrine therapy within 3 months.
5. ECOG performance status 0-2.
6. Adequate bone marrow, liver, renal, and coagulation function as defined in the protocol (ANC ≥1.5×10^9/L, hemoglobin ≥9.0 g/dL, platelets ≥80×10^9/L; TBIL ≤1.5×ULN; AST/ALT/ALP ≤2.5×ULN; albumin ≥30 g/L; creatinine ≤2×ULN or creatinine clearance ≥30 mL/min; INR ≤1.5 in patients not receiving anticoagulation).
7. Patients voluntarily sign informed consent and are willing and able to comply with study procedures.

Exclusion Criteria:

1. History of hypersensitivity or intolerance to any study drugs.
2. mCRPC (metastatic castration-resistant prostate cancer).
3. Oligometastatic mHSPC intended for upfront radical prostatectomy.
4. History of seizure, medications that may lower seizure threshold, or conditions predisposing to seizures (e.g., TIA, stroke, significant head trauma with loss of consciousness requiring hospitalization) within 12 months before starting study treatment.
5. Major surgery within 4 weeks prior to starting study treatment.
6. Significant cardiovascular or cerebrovascular disease within 6 months (e.g., unstable angina, myocardial infarction, NYHA class III or higher heart failure, stroke, clinically significant arrhythmia requiring treatment).
7. Conditions affecting drug intake or absorption (e.g., inability to swallow, chronic diarrhea, intestinal obstruction).
8. Active infection (e.g., HIV positive, HBsAg positive, HCV positive) which in the investigator's opinion may affect safety or efficacy assessment.
9. Other malignancies within the past 3 years, except adequately treated basal cell carcinoma of the skin.
10. Known brain metastases or leptomeningeal disease.
11. Concurrent participation in another interventional clinical trial or receiving other investigational drugs/devices.
12. Poor compliance or inability to adhere to study procedures and follow-up.
13. Any other severe uncontrolled comorbidities (e.g., poorly controlled hypertension, severe diabetes, neurologic or psychiatric disorders) or conditions that may interfere with study conduct or interpretation, as judged by the investigator.

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2025-11-30 (Estimated); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Radiographic Progression-free Survival (rPFS) | From randomization to radiographic progression or death from any cause, whichever occurs first, up to approximately 24 months.
  rPFS will be assessed according to RECIST v1.1 and PCWG3 criteria using PSMA PET/CT, contrast-enhanced CT, MRI, or bone scan. Radiographic progression is defined as the appearance of new lesions or growth of existing measurable disease as per RECIST v1.1, or new bone lesions according to the PCWG3 "2+2" rule

SECONDARY OUTCOMES:
Overall Survival (OS) | From start of systemic therapy to death from any cause, up to the end of follow-up (approximately 24-30 months).
  Time from treatment initiation to death from any cause. Participants alive at last follow-up will be censored.
Biochemical Progression-free Survival (bPFS) | From start of systemic therapy to biochemical progression or death, up to ~24 months.
  Biochemical progression is defined according to ASTRO/AUA joint guideline: a PSA increase of ≥2 ng/mL above the nadir, confirmed by a second consecutive measurement.
PSA Response Rate at 3 and 6 Months | 3 months and 6 months after treatment
  Proportion of patients with PSA decline ≥50% from baseline at 3 months and 6 months after treatment initiation
Conversion Success Rate | At 6 months (and 12 months for supplementary randomization, if applicable)
  Proportion of patients who achieve "conversion success" after 6 months of systemic therapy, defined as PSMA PET/CT showing no metabolically active lesions (all metastases with SUVmax below liver background or blood pool) and fulfilling randomization criteria.
Safety Endpoints | From first dose to 30 days after last dose or last study visit
  Incidence, type, and severity of adverse events (AEs) and serious adverse events (SAEs), graded according to NCI-CTCAE version 5.0, including treatment-emergent AEs, AEs leading to discontinuation, and treatment-related deaths.
Change from Baseline in EORTC QLQ-C30 Score | From baseline to 3, 6, 12, and 24 months after randomization.
  Changes from baseline in health-related quality of life measured by EORTC QLQ-C30 (e.g., Global Health Status/QoL and functional scales).
Change from Baseline in SF-36 Score | From baseline to 3, 6, 12, and 24 months after randomization.
  Changes from baseline in health-related quality of life measured by SF-36 (e.g., PCS and MCS).
Change from Baseline in FACT-G Total Score | From baseline to 3, 6, 12, and 24 months after randomization.
  Changes from baseline in health-related quality of life measured by FACT-G total score.

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kyriakopoulos CE, Chen YH, Carducci MA, Liu G, Jarrard DF, Hahn NM, Shevrin DH, Dreicer R, Hussain M, Eisenberger M, Kohli M, Plimack ER, Vogelzang NJ, Picus J, Cooney MM, Garcia JA, DiPaola RS, Sweeney CJ. Chemohormonal Therapy in Metastatic Hormone-Sensitive Prostate Cancer: Long-Term Survival Analysis of the Randomized Phase III E3805 CHAARTED Trial. J Clin Oncol. 2018 Apr 10;36(11):1080-1087. doi: 10.1200/JCO.2017.75.3657. Epub 2018 Jan 31. PMID 29384722
- [Result] Ost P, Reynders D, Decaestecker K, Fonteyne V, Lumen N, De Bruycker A, Lambert B, Delrue L, Bultijnck R, Claeys T, Goetghebeur E, Villeirs G, De Man K, Ameye F, Billiet I, Joniau S, Vanhaverbeke F, De Meerleer G. Surveillance or Metastasis-Directed Therapy for Oligometastatic Prostate Cancer Recurrence: A Prospective, Randomized, Multicenter Phase II Trial. J Clin Oncol. 2018 Feb 10;36(5):446-453. doi: 10.1200/JCO.2017.75.4853. Epub 2017 Dec 14. PMID 29240541